CLINICAL TRIAL: NCT06998355
Title: BE.Amycon Amyloidosis Data Registry UZ Leuven
Brief Title: BE.Amycon Registry UZ Leuven
Status: Suspended | Type: Observational
Why Stopped: Merged with other trial
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Vlaams Instituut voor Biotechnologie (Unknown)
Responsible Party: Sponsor
Other Study IDs: BE.AMYCON_UZL_WP2_01
Record Dates: First submitted 2025-05-12; First posted 2025-05-31 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Registry — observational data collection

SUMMARY:
The goal of this observational study is to establish database with (limited) personal and health data of patients diagnosed with amyloidosis (any subtype) in order to get better insights on the disease presentation, disease evolution pattern, treatment plans and responses and survival.

DETAILED DESCRIPTION:
With the support of VIB Grand Challenges Program, this project aims to establish the BElgian AMYloidosis CONsortium (BE.AMYCON) by joining forces of VIB researchers, a state-of-the-art diagnostic platform, and clinicians from various disciplines and different institutes. Such a consortium will address patient needs and improve outcomes on many levels.

In this context, a registry of clinical data is a requirement for both improvement of diagnostics as well as fundamental research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Provide consent and sign informed consent form
* Confirmed diagnosis of amyloidosis (any subtype), systemic and/or localised
* Newly diagnosed or in follow-up during the study time-frame (1 JUN 2025 until 31 DEC 2027)

Exclusion Criteria:

* Not able to provide informed consent
* Not willing to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for the study are newly diagnosed amyloidosis patients and amyloidosis patients in follow up at UZ Leuven Gasthuisberg at moment of EC approval.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Participant baseline demographics | Baseline
  Demographic characteristics of amyloidosis participants will be assessed at baseline.
Participant amyloidosis diagnosis information | Baseline
  Disease characteristics will be collected at moment of diagnosis.
Sequence of treatments in participants with amyloidosis | From enrollment of the patient until death, until loss to follow-up or withdrawal of informed consent, whichever comes first, up to 10 years
  Treatment sequences for participants with amyloidosis within routine clinical care will be assessed.

SECONDARY OUTCOMES:
Best Response | From enrollment of the patient until death, until loss to follow-up or withdrawal of informed consent, whichever comes first, up to 10 years
  Documentation of response rates per line of treatment.
Duration of response | From enrollment of the patient until death, until loss to follow-up or withdrawal of informed consent, whichever comes first, up to 10 years
  Duration of response is defined as the time from the date of initial documentation of a response to the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death.
Time to Next Treatment (TTNT) | From enrollment of the patient until death, until loss to follow-up or withdrawal of informed consent, whichever comes first, up to 10 years
  TTNT is defined as the time from the date of initiation of regimen to the initiation of next regimen for each successive therapy received.
Overall Survival (OS) | From enrollment of the patient until death, until loss to follow-up or withdrawal of informed consent, whichever comes first, up to 10 years
  OS is defined as the time from the date of initiation of therapy to the date of death from any cause (or last documented follow-up).
Progression-free survival (PFS) | From enrollment of the patient until death, until loss to follow-up or withdrawal of informed consent, whichever comes first, up to 10 years
  PFS is defined as the time from the date of initiation of therapy to the date of progression or death of any cause, whichever occurs first (or last documented follow-up).

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided